CLINICAL TRIAL: NCT02939196
Title: Comparison of Pain Accompanying the Use of 3.7 mm and 4 mm Office Hysteroscopy in Nullipara: A Randomized Clinical Trial
Brief Title: Pain in Different Office Hysteroscopy Diameter
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Essam Rashad Abdel-Hafeez Othman, Associate Professor, OB-GYN department-principal investigator, Assiut University
Other Study IDs: OH
Record Dates: First submitted 2016-10-18; First posted 2016-10-19 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Pain Associated Office Hysteroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group(A): 2.7 mm rigid hysteroscopy.
  Interventions: Procedure: office hysteroscopy 3.7
- Group(B): 2.9 mm rigid hysteroscopy.
  Interventions: Procedure: office hysteroscopy 4

INTERVENTIONS:
Procedure: office hysteroscopy 3.7 — office hysteroscopy with a 3.7 -mm outer sheath
  Groups: Group(A)
Procedure: office hysteroscopy 4 — office hysteroscopy with a4-mm outer sheath
  Groups: Group(B)

SUMMARY:
The purpose of the investigators'study was To compare 2 different diameter rigid hysteroscopy in vaginoscopic approach regarding pain during and after the procedure.

And to evaluate patient acceptability and tolerability in order to determine the best way to perform hysteroscopy in an outpatient setting.

DETAILED DESCRIPTION:
Office hysteroscopy is used as diagnostic tool to investigate abnormal uterine bleeding and other diseases involving the uterine cavity one of The main limitation to its widespread use is feared from pain and low patient tolerability Narrower diameter hysteroscopy and endometrial biopsy devices are being developed to improve the acceptability of office hysteroscopy. Miniature optical systems allow performance of most diagnostic and operative hysteroscopy (after proper patient selection) in an outpatient or office setting .Flexible hysteroscopy seem to be less painful at the beginning and during the procedure ,but the optical qualities are poor Hysteroscopy is safe, feasible and accurate procedure for diagnosing intrauterine pathology.

Provision of outpatient based diagnostic and operative services are gaining prominence as a standard of cure but the experience of pain can be off-putting for patients having outpatient diagnostic hysteroscopy.

saline solution is an excellent alternative to carbon dioxide in women undergoing outpatient hysteroscopy, and there are fewer complications

ELIGIBILITY:
Inclusion Criteria:

* Woman with nulliparous cervix

Exclusion Criteria:

* Pregnancy.
* female genital cancer
* Active pelvic infection
* Multipara
* patient not receiving misoprostol

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — because hysteroscopy done only in female
Study Population: female patent between 20 to 45 years old who under go office hysteroscopy
Sampling Method: Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-07 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Pain more than 4 (according visual analogue scale | 5 minute

CONTACTS AND LOCATIONS:
Overall Officials: Essam Othman, MD, Principal Investigator — Assiut
Locations (1):
- Essam Othman, Assiut, Cairo, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: No